CLINICAL TRIAL: NCT06725160
Title: Maternal Positive Affect Socialization and Child Neural Reward Response
Brief Title: Parent Encouragement And Coaching of Happiness in Youth
Acronym: PEACHY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Morgan, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY24040170; R01MH135881 (NIH)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Depression; Parent-Child Relations
Keywords: depression; reward; neural; behavior; parent; early childhood
MeSH Terms: conditions — Depression; Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Coaching (Experimental): Parents will receive 3 sessions based on PCIT-ED aimed at increasing child positive affect.
  Interventions: Behavioral: Parent Coaching
- Active Control (Active Comparator): Parents will receive 3 sessions based on traditional PCIT providing more general parenting supporting, including basic psychoeducation and parenting skills.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Parent Coaching — Three sessions of parent coaching of child positive affect will be administered based on modules from PCIT-ED.
  Other Names: PCIT-ED
  Arms: Parent Coaching
Behavioral: Active Control — General parent support and psychoeducation based on components of standard PCIT.
  Arms: Active Control

SUMMARY:
The goal of this mechanistic clinical trial is to examine whether parent-coaching aimed at increasing child positive affect will increase child neural response to reward. The main questions it aims to answer are:

Aim 1. Characterize child neural reward response and its relation to maternal socialization of positive emotions at baseline in healthy young children.

Aim 2. Evaluate how coaching-related changes in maternal socialization of positive emotion expression contribute to increases in child neural reward response over time.

Aim 3. Examine how maternal socialization of positive emotion expression contributes to increases in child neural reward response in the moment.

Participating mother-child dyads will be randomized to either 3 sessions of parent coaching of child positive affect or 3 sessions of a general parenting support intervention and neural response to reward and affective behavior will be examined pre and post intervention.

DETAILED DESCRIPTION:
Reward-related brain function is consistently linked to greater motivation, pleasure, and goal-directed behavior and lower risk for depression across the lifespan. Healthy neural reward response supports socioemotional development, particularly during early childhood as self-regulatory skills and child reward-related brain function are rapidly developing in the context of the caregiving environment. Maternal socialization of positive emotion is one important influence on early reward circuitry development. Mothers with depression are more likely to discourage (and less likely to encourage) child positive emotions compared to healthy mothers, which may contribute to early neural reward alterations in their children. Characterizing mechanisms of influence of maternal socialization on child neural reward response and positive emotion during early childhood is a critical window of opportunity when parents have a large influence on child socioemotional development. Importantly, maternal behavior is amenable to change by training parents on emotion coaching, and these maternal behavior changes may result in direct and immediate changes in child neural reward function. Thus, the overarching aim of this proposal is to use a mechanistic trial design to experimentally test the hypothesis that maternal encouragement of child positive emotion will lead to in-vivo increases in child neural reward response. Event-related potentials (ERPs) are uniquely suited to non-invasively assess in-vivo, fast-occurring changes in child reward response during parent-child interactions, including reward positivity (RewP), and the late positive potential (LPP) amplitudes. Toward this aim, the investigators will randomize 180 mothers with clinically significant depression symptoms and their 4- to 6-year-old children (50% female) to receive either 3 control sessions or 3 positive emotion coaching modules from the Parent-Child Interaction Therapy-Emotion Development (PCIT-ED, which trains mothers on how to encourage positive emotion in their young children. Children will complete reward tasks at pre- and post-coaching, while neural reward response is assessed via ERP (RewP and LPP) with their mothers present allowing for in-vivo assessment of maternal behavior. At both timepoints, the investigators will assess child neural reward response and mothers' self-reported maternal socialization behaviors. Understanding how disrupted neural reward responding develops in early childhood is critical for the promotion of child emotional wellness and can be directly used to develop preventive interventions tailored to young children at familial risk for depression.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* Birth mother (biologically female, any gender)
* Providing regular care for participating child (i.e., at least 50% of time)
* Elevated, clinically significant levels of depression (16 or higher on CES-D)
* Aged 18+

Exclusion Criteria for Mothers:

* Lifetime history of a bipolar disorder
* Lifetime history of a psychotic disorder

Inclusion Criteria for Participating Child:

-Aged 4-6 years

Exclusion Criteria for Participating Child:

* T-score greater than 63 on the internalizing or externalizing composites of the CBCL
* Lifetime history of a psychiatric illness
* Lifetime history of neurodevelopmental disorder
* Lifetime history of neurological disorder

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Reward Positivity (RewP) | From baseline week 1 to final assessment week 5 (week 10 maximum)
  The Reward Positivity (RewP) ERP component of the EEG signal is the mean amplitude (μV; microvolt) on gain-loss trials during receipt of reward related feedback in a computerized reward task with higher RewP amplitudes indicating greater reward response (i.e., more favorable outcome).

SECONDARY OUTCOMES:
Parent Responses to Child Positive affect Scale (PRCPS) | From baseline week 1 to final assessment week 5 (week 10 maximum)
  Change in total score (sum of 7-point Likert scores) on the mother-reported Parent Responses to Child Positive affect Scale (PRCPS) encouragement subscale. The range of possible scores for this outcome is 0 to 84 with higher scores reflecting higher encouragement (i.e., more favorable outcome).
Behavioral Coding of Parental Encouragement of Child Positive Emotion | From baseline week 1 to final assessment week 5 (week 10 maximum)
  Parent and child positive emotion will be coded separately on a 0 - 2 scale in 5 second increments. Parental encouragement of child positive emotion will be calculated as the proportion of epochs in which mothers display positive emotion subsequent to child positive emotion expression in the previous epoch. Higher scores indicate greater parental encouragement of child positive emotion (i.e., more favorable outcome).
Late Positive Potential (LPP) | From baseline week 1 to final assessment week 5 (week 10 maximum)
  The Late Positive Potential (LPP) ERP component of the EEG signal is the mean amplitude (μV; microvolt) on positive-negative trials during a picture viewing computerized task. Great LPP amplitudes to positive vs. neutral pictures indicate greater response to positive affect (i.e., more favorable outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Judith M Morgan, PhD, Principal Investigator — University of Pittsburgh; Lauren M. Bylsma, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the NIH NDA per NIH requirements, which include all primary study measures and demographic information. Participant identifying information is used to create an anonymized GUID to identify participants in the NDA but no identifiable information will be shared publicly.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will begin to upload data to the NIH NDA beginning in July 2025 per NIMH requirements, which would then be made publicly available by November 2025. Data in the NDA will be made available indefinitely as long as the NDA exists as a resource.
Access Criteria: Informed consent documents, protocol information, and statistical analysis plan information will all be uploaded to clinicaltrials.gov. Access to participant level data will be managed by the NIH National Data Archive where all the individual participant data and supporting information will be uploaded. Additional data regarding statistical analyses and corresponding code will be provided as supplemental material to publications that use this data. Since this is a mechanistic clinical trial and not an RCT, a CSR is not applicable.
URL: https://nda.nih.gov/